CLINICAL TRIAL: NCT03416595
Title: A Randomized, Double-blinded, Parallel, Placebo-controlled Study to Investigate the Efficacy of Lb Paracasei [Junlebao Lp. N1115] as a Probiotic to Enhance Gut Development in Young Children
Brief Title: A Study on Efficacy of Feeding N1115 Probiotic Supplement to Young Children
Acronym: N1115Baby
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Junlebao Dairy Group Co., Ltd. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); Teagasc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Lp. N1115 in Young Children
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-01

CONDITIONS: Intestinal Growth of Young Children
Keywords: probiotic; Lactobacillus paracasei N1115; young children

STUDY DESIGN:
Intervention Model Description: The model is a randomized, double-blinded, parallel, placebo-controlled intervention study to assess effect of N1115 Probiotic Supplement (containing Junlebao Lp. N1115) on gut development in young children. Up to 60 healthy children, between the ages of 6 months and 3 years who were born by caesarean section will be recruited into this study. Participants will be randomly assigned to one of two treatment groups, one group is N1115 Probiotic Supplement intervention which contains Lp. N1115 and maltodextrin, the other group is placebo intervention which contains maltodextrin only.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N1115 Probiotic Supplement (Active Comparator): A probiotic supplement containing Lactobacillus paracasei N1115 [Junlebao Lp. N1115] Participators, who met inclusion criteria, will receive following product during 8 weeks: N1115 Probiotic Supplement in the form of powder packaged in sachet (one sachet containing 10^9 CFU Lp. N1115).
  Interventions: Dietary Supplement: N1115 Probiotic Supplement
- Placebo control (Placebo Comparator): Dietary Supplement: Placebo Participators, who met inclusion criteria, will receive an identical N1115 Probiotic Supplement looking and tasting placebo.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: N1115 Probiotic Supplement — Participators will receive a sachet each day during 8 weeks. The contents of the sachet should be added to warm water or milk, mixed until fully dissolved and served within 15 minutes.
  Other Names: Junlebao Lp. N1115
  Arms: N1115 Probiotic Supplement
Dietary Supplement: placebo — Participators will receive a sachet each day during 8 weeks. The contents of the sachet should be added to warm water or milk, mixed until fully dissolved and served within 15 minutes.
  Arms: Placebo control

SUMMARY:
The aim of the study is to examine the intervening effects of N1115 Probiotic Supplement (containing Junlebao Lp. N1115) on gut development in young children at the age of 6 month to 3 years by the way of a randomised, double-blinded, parallel, placebo-controlled clinical trial, and to explore the change of intestinal microbiota composition and healthy condition after intervention.

DETAILED DESCRIPTION:
N1115 Probiotic Supplement contains Lactobacillus paracasei N1115 [Junlebao Lp. N1115], a lactobacillus bacteria strain isolated from traditional homemade yogurt in North China. In recent studys feeding Junlebao Lp. N1115 to C57BL/6 mice, the data suggest that Lp. N1115 enhances intestinal development in neonatal mice, and may confer benefits on the growth at early stage of life.

This study is to investigate if a N1115 Probiotic Supplement product containing Lp. N1115 will improve intestinal health in young children. This randomised, double-blinded, placebo-controlled trial includes two treatment groups which respectively need to recruit 30 volunteers born by cesarean section and aged from 6 months to 3 years. The study group receives N1115 Probiotic Supplement, while the control group receives placebo. The trial lasts for 8 weeks and include four time points of data collection. The stool consistency of children will be recorded everyday, the saliva and stool samples will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 6 months and ≤ 3 years,
2. Child was born by caesarean section,
3. Parent/Guardian has given written informed consent,
4. Be in generally good health as determined by the investigator.

Exclusion Criteria:

1. Are currently taking probiotics or prebiotics, or have taken them in the past 2 weeks,
2. Unwilling to avoid probiotics/prebiotics for the duration of the study,
3. Has any food allergies or an allergy or hypersensitivity to any component of the study products, including, milk proteins allergy or cow's milk allergy,
4. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any condition which contraindicates, in the investigators judgement, entry to the study),
5. Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results,
6. Subjects have taken antibiotics within the past 3 months (history of antibiotic use in previous 6 months recorded),
7. Subjects may not be receiving treatment involving experimental drugs,
8. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.
9. Subjects may not be receiving treatment involving experimental drugs,
10. Exposure to any non-registered drug product within 30 days prior to screening visit.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Defecation improvement | 8 weeks
  Compare the defecation condition of child both in intervention group and placebo group by the way of recording the questionnaire each day.
  Record number of defecation and type of stool based on Bristol Stool Scale.
GI symptoms | 8 weeks
  Compare the gastrointestinal symptoms of child both in intervention group and placebo group by the way of recording the questionnaire each day.
  Record number of flatulence, bloating, cramps and diarrhea compared between child in intervention group and placebo group.

SECONDARY OUTCOMES:
Fecal microbiota | study week 0, 4 and 8
  Analysis diversity of fecal microbiota, using 16S rRNA gene sequencing, both in intervention group and placebo group to study their gut microbiota composition
Salivary cortisol | study week 0, 4 and 8
  Analysis changes in salivary cortisol, using chemiluminescence immunoassay detection, both in intervention group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skillington, Postgraduate, Study Director — The director of this clinical trial in Ireland
Locations (1):
- Atlantia Clinical Food Trials, Cork, Blackrock, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03416595/Prot_000.pdf